CLINICAL TRIAL: NCT03767777
Title: Prospective Study for Aortic Arch Therapy With stENt-graft for Chimney technologY：A Prospective, Multi-center, Objective Performance Criteria Clinical Trial
Brief Title: Prospective Study for Aortic Arch Therapy With stENt-graft for Chimney technologY（PATENCY）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTP84-01
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Aortic Dissection
Keywords: Aortic arch; Aortic disease; Aortic Dissection; Stent Graft
MeSH Terms: conditions — Dissection, Thoracic Aorta; Aortic Diseases; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants will be treated with Artery Stent Graft System Intervention: Device: Artery Stent Graft System
  Interventions: Device: Artery Stent Graft System

INTERVENTIONS:
Device: Artery Stent Graft System — The Artery Stent Graft System consists of Ankura pro Aorta Stent Graft System along with Longuette Aortic Branch Stent Graft System for chimney technique in the aim of revascularization of aorta branches.The Ankura pro aorta stent graft and Longuette Aortic Branch Stent Graft System are pre-assembled within delivery system. During the operation, the stent graft was delivered to the target lesion location of the vascular real cavity through a delivery system, which was accurately positioned and released to isolate the ruptured opening of aortic dissection, block the continuous flow of blood into the false cavity of the dissection, and avoid further tearing or even rupture of the dissection.

SUMMARY:
A prospective, multi-centre, objective performance criteria clinical trial to evaluate the safety and efficacy of Artery Stent Graft System manufactured by Lifetech Scientific (Shenzhen) Co., LTD. for the thoracic aortic dissection involving the aortic arch.

DETAILED DESCRIPTION:
This clinical trial was conducted in a qualified clinical trial institution. Investigators will use Artery Stent Graft System manufactured by Lifetech Scientific (Shenzhen) Co., LTD. to treat patients with thoracic aortic dissection involving the aortic arch. This is a Prospective, Multi-center, Objective Performance Criteria Clinical Trial. It is expected to submit to the ethics committee of the lead unit for review in Sep 2018, and complete the implantation of 150 patients in 18 centres nationwide within 12 months, and interim follow-up was conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery, long-term follow-up will be performed at 24 months postoperatively, 36 months postoperatively, 48 months postoperatively and 60 months postoperatively.

This trial will evaluate whether the device reached the primary safety endpoint and primary efficacy endpoint through two primary endpoint indicators: the incidence of major adverse events (MAE) within 30 days and the success rate of aortic dissection treatment 12 months after surgery.

This trail will evaluate whether the device reached the secondary safety endpoint and efficacy endpoint through several secondary endpoint indicators:

1. the incidence of all-cause death at 30 days, 6 months, 12 months and 2-5 years after surgery
2. the incidence of thoracic aortic dissection-related death at 30 days, 6 months, 12 months and 2-5 years after surgery
3. the incidence of severe adverse events (SAE) at 30 days, 6 months, 12 months and 2-5 years after surgery
4. the incidence of the device-related adverse events (AE) at 30 days, 6 months, 12 months and 2-5 years after surgery
5. the Incidence of left upper limb ischemia at 30 days, 6 months, 12 months and 2-5 years after surgery
6. the incidence of type I or type III leakage at 30 days, 6 months, 12 months after surgery
7. the incidence of graft migration at 30 days, 6 months, 12 months after surgery
8. the branching vascular patency rate at 30 days, 6 months, 12 months after surgery
9. the Incidence of Thoracic aortic dissection -related surgical conversion or re-intervention at 30 days, 6 months, 12 months and 2-5 years after surgery According to the guidelines for clinical trials of aortic stent system, the sponsor will apply for NMPA listing registration after completing a 12-month primary endpoint assessment, and annually follow-up will be conducted until the fifth year for the long-term efficacy observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are 18 years and older, but less than 85 years old and not pregnant or lactating;
2. Patients who can understand the purpose of the trial, voluntarily participate in and sign the informed consent, and are willing to complete the follow-up according to the requirements of the protocol;
3. Patients diagnosed as thoracic aortic dissection involving the arch, and the left subclavian artery branching vessel needs to be revascularized;
4. Aortic proximal landing zone ≥15mm；
5. Aortic proximal diameter in the range of 25-44mm;
6. The left subclavian artery distal landing zone≥15mm;
7. The left subclavian artery diameter in the range of 5-18mm；
8. Patients who have eligible imported arterial vessels.

Exclusion Criteria:

1. Patients with severe stenosis, calcification in the landing area of the stent and easily lead to incomplete stent apposition;
2. Patients need intervention for other vascular diseases (such as coronary artery /renal artery) in the same surgery, or patients with heart disease and medicine treatment will be affected by the intervention；
3. Patients with a history of myocardial infraction or acute coronary syndromes in 3 months；
4. Patients with a history of cerebrovascular events or gastrointestinal bleeding in 3 months, antiplatelet agent and anticoagulant contraindication, or tendency of hemorrhage；
5. Patients have received any major surgical or interventional therapy within 30 days (Operation Classification reaches III or above) or have received interventional therapy;
6. Patients will receive any major selective operation or interventional therapy in 30days (Operation Classification reaches III or above) or will received interventional therapy;
7. Patients already treated with an thoracic aortic stent graft and the stent graft can affect operation or intersection part existing between the graft covering area；
8. Patients with genetic connective tissue disease (e.g., Marfans syndrome) or aorta hereditary disease；
9. Patients with infectious aortic dissection;
10. Patients with acute systemic infection;
11. Patients with major organ failure or other serious diseases;
12. Patients with a history of active bleeding, clotting disorder, or rejection of blood transfusions;
13. Patients with liver dysfunction: preoperative creatinine was 2.5 times higher than the normal upper limit; Alanine transaminase (ALT) or Aspartate transaminase (AST) were 5 times higher than the normal upper limit; serum total bilirubin (STB) was 2 times higher than the normal upper limit;
14. Pregnant or lactating women or women who plan to get pregnant;
15. Patients who can not tolerate to Anaesthetic；
16. Patients with a history of allergy to contrast media, stents and conveyor materials (including nickel and titanium, polyester, PTFE, and nylon polymer materials);
17. Patients with a life expectancy less than 12 months（such as terminal malignant tumor）；
18. Patients who were not suitable for endovascular treatment, judged by the investigator;
19. Patients who participated in clinical trials of other drugs or medical devices at the same time.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The treatment success rate of aortic dissection at 12 months post-implant | 12 months after surgery
  Assessment of the rate of successful disease treatment defined as immediate technical success and freedom from secondary intervention at 12 months of follow-up.
  Technique success means delivery system is successfully transported to the predetermined position, both of aorta stent graft and aortic branch stent graft successfully expanded and delivery system withdraw successfully.No type I/III endoleak at the end of operation, no conversion to open surgery. (Adjuvant Interventions during operation do not defined as technical failure.)
Incidence of no major adverse events (MAE) occurred at 30 days post-implant | 30 days after surgery
  Major Adverse events (MAE) are defined as aortic dissection related mortality, ischemic stroke, and paraplegia.

SECONDARY OUTCOMES:
Incidence of all-cause death | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of Aortic dissection dissection-related death | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of Serious Major Adverse Event（SAE） | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of device related adverse events（AE） | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of left upper limb ischemia | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of I/III type endoleaks | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of graft migration | 30 days，6 months, 12 months and 2-5 years after surgery
Branching vascular patency rate | 30 days，6 months, 12 months and 2-5 years after surgery
Incidence of Thoracic aortic dissection -related surgical conversion or re-intervention | 30 days，6 months, 12 months and 2-5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chang Shu, professor, Principal Investigator — Central South University
Locations (21):
- China (21):
  - Fuwai hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospita, Beijing, Beijing Municipality
  - The Frist Hospital of Lanzhou University, Lanzhou, Gansu
  - LIU ZHOU WORKER'S HOSPITAL,Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - The second affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital,Tongji Medical College of Huazhong University of Science&Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital (Nanjing Gulou Yi Yuan), the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The first affiliated hospital of soochow university, Suzhou, Jiangsu
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - West China hospital of sichuan university, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjing Medical University General Hospital, Tianjin, Tianjin Municipality
  - The first people's hospital of yunnan province, Kunming, Yunnan

REFERENCES:
- [Derived] Shu C, Wan Z, Luo M, Fang K, Hu J, Zuo J, Li X, Li Q, He H, Li X. Mid-term results of a prospective study for aortic dissection with a gutter-plugging chimney stent graft. Eur J Cardiothorac Surg. 2024 May 3;65(5):ezae135. doi: 10.1093/ejcts/ezae135. PMID 38569918
- [Derived] Liu Y, Fang K, Luo MY, Xiao ZH, Yang P, Lu C, Zhang Y, Wang HY, Xie Y, Xu ZY, Zhang HW, Shu C, Hu J. Single-Center Preliminary Experience with Gutter-Plugging Chimney Stent-Graft for Aortic Dissection. Cardiovasc Intervent Radiol. 2023 Jun;46(6):703-712. doi: 10.1007/s00270-023-03444-8. Epub 2023 May 17. PMID 37198293